CLINICAL TRIAL: NCT04507425
Title: High Flow Nasal Cannula With Noninvasive Ventilation and Its Effect on High Risk Trauma Patients
Brief Title: High Flow Nasal Cannula With Noninvasive Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12248
Record Dates: First submitted 2020-07-25; First posted 2020-08-11 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Acute Respiratory Failure
Keywords: acute respiratory failure; mechanical ventilation
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into 1 of 3 interventions: nasal cannula, high flow nasal cannula, and high flow nasal cannula plus noninvasive ventilation within each of two groups: patients admitted to ICU without being intubated OR intubated patients undergoing an extubation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Not Intubated (Active Comparator): Patients admitted with a trauma injury who do not need to be intubated to receive treatment. Intubated means putting a tube down your throat to keep your airway from collapsing. Participants will be randomized to receive one of the three interventions in this arm.
  Interventions: Other: Standard of Care - Nasal Cannula; Other: High-flow nasal cannula; Other: HFNC plus non-invasive ventilation
- Intubated Patients Undergoing Extubation (Active Comparator): Patients admitted with a trauma injury who had to be intubated for treatment of their injury. Interventions administered after the tube is extubated (removed from throat). Participants will be randomized to receive one of the three interventions in this arm.
  Interventions: Other: Standard of Care - Nasal Cannula; Other: High-flow nasal cannula; Other: HFNC plus non-invasive ventilation

INTERVENTIONS:
Other: Standard of Care - Nasal Cannula — Standard of care. Flexible tube to provide extra oxygen when patients need a little help, but are not in respiratory distress.
Other: High-flow nasal cannula — Same as nasal cannula, except the oxygen is heated or humidified and the flow is stronger, pushing air into the lungs to help keep the airway open.
  Other Names: HFNC
Other: HFNC plus non-invasive ventilation — This method uses HFNC as described above and adds noninvasive ventilation which is similar to CPAP machine and uses a mask rather than having to intubate (putting a tube down your throat to keep your airway from collapsing).

SUMMARY:
This is a prospective, randomized, unblinded trial of trauma patients in the ICU who are identified as being at a high risk to develop acute respiratory failure.

We hope that this study will help the study team to identify how best to use a more aggressive respiratory treatment strategy in a high risk trauma population (thoracic trauma or trauma patients requiring thoracic surgery, spine surgery, or open abdominal procedures) to try and decrease the need for intubation with mechanical ventilation.

DETAILED DESCRIPTION:
All patients consented will be randomly assigned into one of three groups: nasal cannula (control group, our current standard of care), high-flow nasal cannula, high-flow nasal cannula plus noninvasive ventilation.

After obtaining consent, patient will be randomized to interventions 1:1:1 within each of two groups: patients admitted to the ICU without being intubated OR intubated patients undergoing an extubation.

Randomization will be managed through RedCap. After consent, the treating clinician will log into RedCap to obtain the patient's treating assignment.

The primary outcome of interest is failure of conservative ventilation intervention in prevention of initial intubation or prevention of reintubation.

A chart review of all enrolled patients will be done quarterly to assess morbidity, mortality, and outcomes.

No placebo will be used as all qualifying patients will be placed on nasal cannula, high-flow nasal cannula, or high-flow nasal cannula plus noninvasive ventilation. All other treatments will be standard of care.

Participants in the study will continue until the patient is discharged from the trauma ICU.

The study will end when the last person enrolled has been discharged from the trauma ICU. If patient's participation ends prematurely, available data will be entered into the database and evaluated appropriately.

This study will take place at the OU Medical Center (OUMC) among patients admitted to the Trauma Intensive Care Unit.

Consent for study enrollment will take place at OUMC during discussion with physician providing trauma care and the patient, family member, or next of kin consenting for the study.

The following data will be collected and recorded: Supplemental oxygen requirements, Date/Time of arrival, Date/Time of Admission to ICU, Date/Time of intubation procedure, Date/Time of extubation, Ventilator settings, Duration of intubation, Comorbidities, PaCO2 values, PaO2 values, Vital signs at arrival and at admission to ICU, Age,Gender, Weight, Height, BMI, Traumatic injuries, Diagnosis, Past medical history/medical co-morbidities, Glasgow coma scale, Oxygen saturation, Negative inspiratory force score, Rapid shallow breathing index score, Pulmonary treatments, including an intolerance to therapy, Injury Severity Score (ISS) and/or Abbreviated Injury Scale (AIS).

ELIGIBILITY:
Inclusion Criteria:

1. Adults at least 18 years of age
2. Admission to an intensive care unit by the trauma surgery service
3. Trauma patients receiving any respiratory therapies
4. High risk patients, including intubation, post-operative, chronic cardiac or pulmonary comorbidities
5. Thoracic injuries, including rib fractures, sternal fractures, spinal fractures, pulmonary contusions, pneumothorax, hemothorax, diaphragm injury
6. Postoperative from thoracic surgery
7. Postoperative from spine surgery in patients without spinal cord injury
8. Abdominal injuries requiring open abdominal surgery
9. No contraindications to using high flow nasal cannula or noninvasive ventilation

Exclusion Criteria:

1. Contraindication to using high flow nasal cannula or noninvasive ventilation
2. Intolerance of pulmonary therapies
3. No one able to give informed consent
4. Long-term treatment with noninvasive ventilation prior to hospital admission
5. "Do not intubate" order at time of extubation
6. Unplanned extubation (accidental or self-extubation)
7. Age < 18 years of age
8. Traumatic brain injury with GCS < 8
9. Spinal cord injury
10. Chronic neuromuscular disease
11. Sinus precautions due to facial/sinus fractures

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
failure rates-nonintubated patients | first 48 hours
  Among injured patients admitted to the intensive care unit (ICU) without being intubated, do failure rates within the first 48 hours of ICU admission differ with respect to type of initial respiratory intervention: nasal cannula, high-flow nasal cannula (HFNC), or HFNC plus non-invasive ventilation (BiPAP). Failure is defined as escalation to intubation.
failure rates-intubated patients | first 48 hours
  Among injured patients arriving intubated or who undergo intervention after hospital arrival, do failure rates within the first 48 hours after extubation differ with respect to type of initial respiratory intervention: nasal cannula, high-flow nasal cannula (HFNC), or HFNC plus non-invasive ventilation (BiPAP). Failure is defined as requiring reintubation.

SECONDARY OUTCOMES:
Mortality | Up to 2 years
  Assess mortality of enrolled patients by quarterly retrospective chart reviews.
Length of hospital stay | up to 60 days
  Compare length of hospitalization between groups
Length of ICU stay | up to 30 days
  Compare length of ICU stay between groups
Discharge location | up to 60 days
  was patient discharged to home, rehabilitation facility, skilled nursing, death; compare between groups
Complications | up to 2 years
  Compare complications (such as need to be mechanically ventilated, infections, etc.) between groups

CONTACTS AND LOCATIONS:
Overall Officials: Celia Y Quang, MD, Principal Investigator — University of Oklahoma
Locations (1):
- OU Medical Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Thille AW, Boissier F, Ben-Ghezala H, Razazi K, Mekontso-Dessap A, Brun-Buisson C, Brochard L. Easily identified at-risk patients for extubation failure may benefit from noninvasive ventilation: a prospective before-after study. Crit Care. 2016 Feb 26;20:48. doi: 10.1186/s13054-016-1228-2. PMID 26926168
- [Result] Thille AW, Muller G, Gacouin A, Coudroy R, Decavele M, Sonneville R, Beloncle F, Girault C, Dangers L, Lautrette A, Cabasson S, Rouze A, Vivier E, Le Meur A, Ricard JD, Razazi K, Barberet G, Lebert C, Ehrmann S, Sabatier C, Bourenne J, Pradel G, Bailly P, Terzi N, Dellamonica J, Lacave G, Danin PE, Nanadoumgar H, Gibelin A, Zanre L, Deye N, Demoule A, Maamar A, Nay MA, Robert R, Ragot S, Frat JP; HIGH-WEAN Study Group and the REVA Research Network. Effect of Postextubation High-Flow Nasal Oxygen With Noninvasive Ventilation vs High-Flow Nasal Oxygen Alone on Reintubation Among Patients at High Risk of Extubation Failure: A Randomized Clinical Trial. JAMA. 2019 Oct 15;322(15):1465-1475. doi: 10.1001/jama.2019.14901. PMID 31577036
- [Result] Xu Z, Li Y, Zhou J, Li X, Huang Y, Liu X, Burns KEA, Zhong N, Zhang H. High-flow nasal cannula in adults with acute respiratory failure and after extubation: a systematic review and meta-analysis. Respir Res. 2018 Oct 16;19(1):202. doi: 10.1186/s12931-018-0908-7. PMID 30326893
- [Result] Honrubia T, Garcia Lopez FJ, Franco N, Mas M, Guevara M, Daguerre M, Alia I, Algora A, Galdos P. Noninvasive vs conventional mechanical ventilation in acute respiratory failure: a multicenter, randomized controlled trial. Chest. 2005 Dec;128(6):3916-24. doi: 10.1378/chest.128.6.3916. PMID 16354864
- [Result] Halub ME, Spilman SK, Gaunt KA, Lamb KD, Jackson JA, Oetting TW, Sahr SM. High-flow nasal cannula therapy for patients with blunt thoracic injury: A retrospective study. Can J Respir Ther. 2016 Fall;52(4):110-113. Epub 2016 Nov 1. PMID 30996619
- [Result] Gaunt KA, Spilman SK, Halub ME, Jackson JA, Lamb KD, Sahr SM. High-Flow Nasal Cannula in a Mixed Adult ICU. Respir Care. 2015 Oct;60(10):1383-9. doi: 10.4187/respcare.04016. Epub 2015 Jun 9. PMID 26060320
- [Result] Lamb KD, Spilman SK, Oetting TW, Jackson JA, Trump MW, Sahr SM. Proactive Use of High-Flow Nasal Cannula With Critically Ill Subjects. Respir Care. 2018 Mar;63(3):259-266. doi: 10.4187/respcare.05793. Epub 2017 Dec 5. PMID 29208754